CLINICAL TRIAL: NCT02414243
Title: A Multicenter, Randomized, Controlled, Cross-over Study to Assess Hypoallergenicity of a New Amino-acid Based Infant Formula in Children With Cow's Milk Allergy
Brief Title: Study to Assess Hypoallergenicity of a New Amino-acid Based Infant Formula in Children With Cow's Milk Allergy
Acronym: RAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Ordesa (Industry)
Collaborators: OPBG Clinical & Research Services S.R.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: RAF-01-015
Record Dates: First submitted 2015-02-11; First posted 2015-04-10 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- New Amino Acid formula (Experimental): New Amino-Acid based Infant Formula
  Interventions: Other: New Amino Acid formula
- Control formula (Active Comparator): Commercially available Amino Acid Formula
  Interventions: Other: Commercially available Amino Acid Formula

INTERVENTIONS:
Other: New Amino Acid formula — Ordesa's Amino-Acid based Infant Formula
  Arms: New Amino Acid formula
Other: Commercially available Amino Acid Formula — Commercially available Amino Acid Formula
  Arms: Control formula

SUMMARY:
This is a prospective, controlled, multi-country study to verifying the hypoallergenicity of the new amino acid-based formula in infants and children aged< 12 years with documented cow's milk protein allergy (CMPA).

DETAILED DESCRIPTION:
Not Provided

ELIGIBILITY:
Inclusion Criteria:

* Children with documented cow's milk allergy, confirmed by one of the following criteria, within six months prior to study start (visit 2):

  * Positive double-blind, placebo-controlled oral food challenge (DBPCFC) with cow's milk OR
  * Positive open or single-blind oral food challenge with cow's milk carried out under the supervision of a specialist in children with clear immediate reactions and a positive test for specific IgE (in serum [sIgE>0,35 KUI/L] or skin prick test [SPT ≥ 3 mm]) OR
  * Reported convincing allergic symptoms following an exposure to milk or a milk-containing food product and detectable serum milk-specific IgE or positive skin prick test
* Aged ≤12 years of age at screening.
* Expected consumption of a minimum of 250ml of study formula per day during the open challenge.
* Written informed consent from one or both parents (depending on the local legislation) or legal representative.

Exclusion Criteria:

* Children who receive breastfeeding at study enrolment.
* Had any chronic medical diseases, chromosomal or major congenital anomalies, or major gastrointestinal disease/abnormalities (other the CMPA); had immunodeficiency; antihistamine [excluding eye drops] use in 7 days prior to a food challenge or oral steroid use within 14 days prior to enrolment; unstable asthma; severe uncontrolled eczema;
* Severe anaphylactic reaction [required ≥ 2 doses of epinephrine] to milk or breast milk within the past 2 years;
* Existing illness that could interfere with formula acceptance or identification of allergic reactions.
* Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements.
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Banzato, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata, Verona, Italy; Maria Pedrosa, MD, Principal Investigator — Hospital Universitario La Paz; Elena Alonso, MD, Principal Investigator — Hospital General Universitario Gregorio Marañón, Madrid, Spain; Montserrat Bosque, MD, Principal Investigator — Hospital Universitario Parc Taulí Sabadell, Barcelona, Spain; Anna Mª Plaza, MD, Principal Investigator — Hospital Sant Joan de Déu, Barcelona, Spain
Locations (1):
- Ospedale Pediatrico Bambino Gesù, Rome, Italy

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765

RESULTS

PARTICIPANT FLOW:
Groups:
- New Amino Acid Formula + Control Formula: New Amino-Acid based Infant Formula and then control formula and then open challenge with new amino acid formula
  New Amino Acid formula: Ordesa's Amino-Acid based Infant Formula
- Control Formula + New Amino Acid Formula: Commercially available Amino Acid Formula + New Amino Acid formula + open challenge with newm formula
  Commercially available Amino Acid Formula: Commercially available Amino Acid Formula
Period: Overall Study
Arm/Group | New Amino Acid Formula + Control Formula | Control Formula + New Amino Acid Formula
Started (41 randomized but 1 patient left study after randomization) | 19 | 21
Moved to the Other Group | 17 | 20
Entered Open Challenge at Home | 17 | 20
Completed | 13 | 17
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Population: 41 patients randomized but 2 patients withdrew before treatment. 39 patients analyzed.
Groups:
- New Aminoacid Formula + Control: Patients that followed the sequence: New aminoacid formula + control formula
- Control Formula + New Aminoacid Formula: Patients that followed the sequence: control formula + new aminoacid formula
- Total: Total of all reporting groups
Arm/Group | New Aminoacid Formula + Control | Control Formula + New Aminoacid Formula | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.43 (2.78) | 1.78 (2.27) | 2.1 (2.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 11 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black | 0 | 1 | 1
  Caucasian | 17 | 17 | 34
  Hispanic | 0 | 1 | 1
  Not Specified | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Italy | 14 | 13 | 27
  Spain | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Hypoallergenicity as Assessed by Reaction to Amino-acid Based Infant Formula
Description: To demonstrate that the test formula does not cause immediate and/or delayed allergic reactions to a double blind placebo control food challenge (DBPCFC) and/or a subsequent open food challenge (OFC). Incidence of immediate and/or delayed allergic reactions to the DBPCFC with the study product and/or active comparator and/or during the subsequent OPEN challenge phase of the study.
Time Frame: 14 days
Population: 41 subjects were enrolled and randomized to formula sequence. Only 30 subjects completed the Open Challenge with SanorE formula.
Measure: Count of Participants; unit: Participants
Groups:
- DBPCFC (New Milk SanorE): DBPCFC: Double blind placebo controlled food challenge (New milk)
- DBPCFC (Control Milk Neocate): DBPCFC: Double blind placebo controlled food challenge (control milk)
- Open Challenge With SanorE: Open challenge with SanorE phase
Arm/Group | DBPCFC (New Milk SanorE) | DBPCFC (Control Milk Neocate) | Open Challenge With SanorE
Number analyzed (Participants) | 30 | 30 | 30
Participants
  Positive | 0 | 0 | 0
  Negative | 30 | 30 | 30
  Inconclusive | 0 | 0 | 0

2. Secondary Outcome: Cow's Milk Allergy Related Symptoms
Description: Cow's Milk Allergy related Symptoms recorded at visit 1 and visit 4 using the Vandenplas symptom-based score (SBS).
  The scoring ranges from 0 to 33. Each symptom has a maximal score of 6, except respiratory symptoms where the maximal score is 3. If final score ≥ 12, the symptoms are likely cow's milk related. This could potentially be CMPA.
  If final score <12, the symptoms are less likely related to cow's milk. Look for other causes.
Time Frame: 14 days
Population: 41 patients randomized but 30 completed. Results are presented as total score summary . It compares changes between visit 4 and visit 1, and comparison were performed globally. No other result available.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Global: Cow's Milk Allergy related Symptoms (Vandenplas)
Arm/Group | Global
Number analyzed (Participants) | 30
score on a scale
  V1 Screening | 1.37 (1.59)
  V4 week 2: number analyzed (Participants) | 29
  V4 week 2 | 0.79 (1.21)

ADVERSE EVENTS:
Time Frame: From screening visit to week 2
Description: In this study, patients received the two treatments, with the sequence A: New aminoacid formula + control formula; or sequence B: control formula + new aminoacid formula. As all patients received the two treatments, adverse events table does not difference between groups and shows global study population.
  There were no serious or non-serious adverse events related to the study treatment reported in this study.
Groups:
- Global: Data from all participants in the study. Data has been presented globally in the final report, no results from different groups. Only occurrence of adverse events.
Arm/Group | Global
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 1/39
Other Adverse Events (participants affected / at risk) | 9/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global (N=39)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Global (N=39)
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Pyrexia (Gastrointestinal disorders) | 4
Asthma (Immune system disorders) | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No